CLINICAL TRIAL: NCT01423812
Title: DRIVESHAFT: Phase IV Randomized, Open-Label Study in HIV-1 Virologically-suppressed Patients On Regimens With Darunavir 600mg/Ritonavir 100mg Twice-daily Switching to Darunavir 800mg/Ritonavir 100mg Once-daily Vs. Continuing Twice-daily Darunavir/Ritonavir Regimens
Brief Title: DRIVESHAFT: Darunavir/Ritonavir In HIV-infected Virologically-suppressed Experienced Subjects
Acronym: DRIVESHAFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruth M. Rothstein CORE Center (Other)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Principal Investigator, Gregory Huhn, Attending Physician, Ruth M. Rothstein CORE Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC114HIV4063
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: HIV
Keywords: HIV; treatment-experienced; protease inhibitor; adherence; lipids
MeSH Terms: interventions — Ritonavir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once-daily Darunavir and ritonavir (Experimental): Subjects switched from Darunavir 600mg plus Ritonavir 100mg twice-daily to Darunavir 800mg plus Ritonavir 100mg once-daily
  Interventions: Drug: Once-daily combination Darunavir and ritonavir
- Twice-daily Darunavir and ritonavir (Active Comparator): Subjects remain on regimens containing Darunavir 600mg plus Ritonavir 100mg twice-daily
  Interventions: Drug: Twice-daily combination Darunavir and ritonavir

INTERVENTIONS:
Drug: Twice-daily combination Darunavir and ritonavir — Subjects randomized 1:1 to remain on regimens containing combination Darunavir 600mg plus Ritonavir 100mg twice-daily
  Other Names: Prezista and norvir twice-daily
  Arms: Twice-daily Darunavir and ritonavir
Drug: Once-daily combination Darunavir and ritonavir — Subjects randomized 1:1 to switch to from combination Darunavir 600mg plus Ritonavir 100mg twice-daily at baseline to the experimental combination Darunavir 800mg plus Ritonavir 100mg once-daily for 48 weeks
  Other Names: Prezista and norvir once-daily
  Arms: Once-daily Darunavir and ritonavir

SUMMARY:
Darunavir is a nonpeptidic protease inhibitor with a high genetic barrier to resistance that evolved from a prototype compound synthesized using structure-based design strategies. Once-daily darunavir at 800mg boosted with 100mg of ritonavir is an effective antiretroviral agent indicated for HIV-infected treatment-naïve patients. In treatment-experienced patients, darunavir was initially approved for twice-daily administration boosted with twice-daily ritonavir at 600mg and 100mg, respectively. Recently, once-daily darunavir/ritonavir was approved for use in treatment-experienced adult patients with viremia with no darunavir resistance mutations. In treatment-experienced patients with viral suppression, switching from an antiretroviral taken twice-daily to a once-daily dose is an attractive option to promote greater patient acceptability and adherence, and potentially minimize side effects and toxicities. Because of darunavir/ritonavir's high genetic barrier to resistance and well-established safety profile at a once-daily dose, switching patients with virologic suppression from twice-daily darunavir/ritonavir to once-daily darunavir/ritonavir will likely confer attributes more favorable to patients through a simplified dosing schedule and lower potential for lipid elevation without the loss of virologic control. DRIVESHAFT is a 48-week Phase 4, randomized, open label, comparative study. The study will be conducted in 60 HIV-1 infected, antiretroviral experienced, virologically-suppressed patients on regimens containing darunavir 600mg/ ritonavir 100mg twice-daily and a minimum of two other antiretrovirals, with a history of 0-1 darunavir-associated resistance mutations. Subjects will be randomized 1:1 to switch to darunavir 800mg/ ritonavir 100mg once-daily or continue on their current regimen. Rates of virologic suppression of once-daily darunavir/ritonavir regimens relative to darunavir/ritonavir twice-daily regimens will be compared, and safety, change from baseline fasting lipid parameters, and adherence will be evaluated.

DETAILED DESCRIPTION:
The Darunavir/Ritonavir In Virologically-suppressed Experienced Subjects Halving an Antiretroviral by Finetuning Therapy (DRIVESHAFT) study was a prospective, randomized, single-centre, two-arm, open-label 48-week pilot study. The aim of DRIVESHAFT was to evaluate the safety and efficacy of switching the DRV/r component from twice-daily to once-daily 800/100 mg compared with those remaining on current therapy among HIV-1-infected, treatment-experienced patients with 0-1 DRV RAMs on a stable regimen including twice-daily DRV/r 600/100 mg. The study was conducted at The Ruth M Rothstein CORE Center (Chicago, IL, USA). The sample size was determined upon feasibility as a single-site study and not powered for non-inferiority. Study enrolment was planned for 60 participants randomized 1:1 to one of two arms: the switch arm from DRV/r 600/100 mg twice daily to DRV/r 800/100 mg once/daily plus current ARV regimen including a minimum of two other agents or remain on current ARV regimen with minimum of three agents inclusive of twice-daily DRV/r. Two DRV 400 mg tablets were used in the once-daily DRV/r arm, with DRV 600 mg tablets administered in the twice-daily DRV/r arm.

DRIVESHAFT inclusion criteria included HIV-1-infected adult (>18 years of age), HIV-1 RNA measurements <40 copies/ml (using a local assay) over at least 12 weeks on a stable regimen including DRV/r 600/100 mg twice daily plus a minimum of two other ARVs, screening HIV-1 RNA<40 copies/ml, have undergone genotypic testing at any time prior to starting current antiretroviral therapy (ART) with evidence of <2 cumulative DRV RAMs, CD4+ T-cell count >50 cells/mm3, and a negative serum pregnancy test at screening visit Participants who were randomized and received at least one dose of study medication were included in efficacy analysis, and the primary end point was the proportion of participants with HIV-1 RNA<40 copies/ml at week 48.

ELIGIBILITY:
Inclusion Criteria:

1. ART-experienced, HIV-1 infected subjects ≥18 years of age.
2. A female subject is eligible to enter and participate in the study if she:

   1. is of non-childbearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy, or bilateral oophorectomy or,
   2. is of child-bearing potential, with a negative pregnancy test at both Screen and Day 1 and agrees to one of the following methods of contraception to avoid pregnancy:

      * Complete abstinence from intercourse from 2 weeks prior to administration of study medications, throughout the study, and for at least 2 weeks after discontinuation of all study medications.
      * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide).
      * Approved hormonal contraception may be administered with darunavir/ritonavir
      * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year
      * Any other method with published data showing that the expected failure rate is <1% per year.

   Any contraception method must be used consistently and in accordance with the approved product label. All subjects participating in the study should be counseled on safer sexual practices including the use of effective barrier methods (e.g. male condom/spermicide).
3. CD4 >50 cells/mm3
4. HIV-1 RNA concentrations at undetectable levels (according to local assay being used) for at least 12 weeks on stable current regimen
5. Current regimen includes darunavir/ritonavir 600/100 mg twice-daily plus a minimum of two other antiretrovirals
6. Negative serum pregnancy test at screening visit

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Known hypersensitivity reaction to agents being utilized in the study
2. >1 cumulative darunavir associated mutations (V11I, V32I, L33F, I47V, I50V, I54L or M, T74P, L76V, I84V, or L89V) detected from any previous genotype or a VircoTYPE HIV-1 darunavir fold-change >10.0 on any previous virtual phenotype
3. Pregnant or breast feeding woman
4. Liver dysfunction with Child-Pugh class C disease or decompensated cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GREGORY G HUHN, MD, Principal Investigator — The Ruth M. Rothstein CORE Center
Locations (1):
- Ruth M. Rothstein CORE Center, Chicago, Illinois, United States

REFERENCES:
- [Background] 1. De Meyer S, et al. Antiviral activity of TMC 114, a potent next generation protease inhibitor against more than 4000 recent recombinant clinical isolates exhibiting a wide range of protease inhibitor resistance profile. Antiviral Ther 2003;8:3S19. 2. De Meyer SD, et al. Phenotypic and genotypic determinants of resistance to TMC 114: pooled analysis of POWER 1,2, and 3. Antiviral Ther 2006;11:S83. 3. Panel on Antiretroviral Guidelines for Adults and Adolescents. Department of Health and Human Services. December 1,2009;1-161. Accessed September 15, 2010. 4. Cahn PK, et al. Efficacy and Safety at 48 Weeks of Once-daily vs Twice-daily DRV.r in Treatment-experienced HIV-1-positive Patients with No DRV Resistance-associated Mutations: The ODIN Trial. Abstract 57. 17th CROI 2010. 5. Moltó J, et al. Treatment simplification to once daily darunavir/ritonavir guided by the darunavir inhibitory quotient in heavily pretreated HIV-infected patients. Antivir Ther. 2010;15(2):219-25.
- [Derived] Huhn GD, Sigman A, Livak B. Simplification from twice-daily to once-daily darunavir/ritonavir in a randomized trial among HIV-infected persons with HIV-1 RNA suppression on antiretroviral therapy. Antivir Ther. 2015;20(8):849-54. doi: 10.3851/IMP2962. Epub 2015 Apr 17. PMID 25881614
- See also: published results — http://www.ncbi.nlm.nih.gov/pubmed/25881614

RESULTS

PARTICIPANT FLOW:
Groups:
- Once-daily Darunavir/Ritonavir: Subjects switched from Darunavir 600mg plus Ritonavir 100mg twice-daily to Darunavir 800mg plus Ritonavir 100mg once-daily
  Once-daily Darunavir/ritonavir: Subjects switched from Darunavir 600mg plus Ritonavir 100mg twice-daily at baseline to Darunavir 800mg plus Ritonavir 100mg once-daily for 48 weeks
- Twice-daily Darunavir/Ritonavir: Subjects remain on regimens containing Darunavir 600mg plus Ritonavir 100mg twice-daily
  Twice-daily Darunavir/ritonavir: Subjects remain on regimens containing Darunavir 600mg plus Ritonavir 100mg twice-daily
Period: Overall Study
Arm/Group | Once-daily Darunavir/Ritonavir | Twice-daily Darunavir/Ritonavir
Started | 30 | 30
Completed | 27 | 26
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Once-daily Darunavir/Ritonavir | Twice-daily Darunavir/Ritonavir | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 48 [36 to 65] | 49 [38 to 66] | 48 [36 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 24 | 25 | 49
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint for Virologic Suppression in HIV-infected Subjects
Description: Proportion of subjects with plasma HIV-1 RNA <40 c/mL at Week 48 using a Missing, Switch, or Discontinuation = Failure (MSDF) algorithm as codified by the FDA's "snapshot" algorithm
Time Frame: 48 weeks after randomization to study medication
Measure: Number; unit: participants
Arm/Group | Once-daily Darunavir/Ritonavir | Twice-daily Darunavir/Ritonavir
Number analyzed (Participants) | 30 | 30
participants | 27 | 25

2. Secondary Outcome: Secondary Efficacy Endpoints
Description: •Proportion of subjects with plasma HIV-1 RNA >200 c/mL at Week 24
Time Frame: Within 24 weeks after randomization to study medication
Population: Population for outcome of subjects with plasma HIV-1 RNA >200 copies/ML at week 24
Measure: Count of Participants; unit: Participants
Groups:
- Once-daily Darunavir and Ritonavir: Subjects switched from Darunavir 600mg plus Ritonavir 100mg twice-daily to Darunavir 800mg plus Ritonavir 100mg once-daily
  Once-daily Darunavir and ritonavir: Subjects switched from Darunavir 600mg plus Ritonavir 100mg twice-daily at baseline to Darunavir 800mg plus Ritonavir 100mg once-daily for 48 weeks
- Twice-daily Darunavir and Ritonavir: Subjects remain on regimens containing Darunavir 600mg plus Ritonavir 100mg twice-daily
  Twice-daily Darunavir and ritonavir: Subjects remain on regimens containing Darunavir 600mg plus Ritonavir 100mg twice-daily
Arm/Group | Once-daily Darunavir and Ritonavir | Twice-daily Darunavir and Ritonavir
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

3. Secondary Outcome: Change in Total Cholesterol From Baseline to 48 Weeks
Description: Absolute change in lipid parameter (total cholesterol mg/dl) of once-daily versus twice-daily darunavir/ritonavir containing regimens over 48 weeks
Time Frame: Within 48 weeks of randomization baseline to study medications
Population: Mean within person change in total cholesterol mg/dl from baseline
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Once-daily Darunavir and Ritonavir | Twice-daily Darunavir and Ritonavir
Number analyzed (Participants) | 30 | 30
mg/dl | -14.2 (0.148) | -3.8 (0.148)
Statistical Analysis 1: Comparison: Once-daily Darunavir and Ritonavir vs Twice-daily Darunavir and Ritonavir; p value; Test type: Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Absolute Value Change in CD4+ From Baseline to Week 48
Description: Absolute value increase in CD4+ cells/mm3 from baseline to week 48
Time Frame: 48 weeks after randomization baseline to study medications
Population: Population for outcome of subjects measuring absolute change in CD4+ at week 48
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | Once-daily Darunavir and Ritonavir | Twice-daily Darunavir and Ritonavir
Number analyzed (Participants) | 30 | 30
cells/mm3 | 19 (0.592) | 39 (0.592)
Statistical Analysis 1: Comparison: Once-daily Darunavir and Ritonavir vs Twice-daily Darunavir and Ritonavir; Test type: Other; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Assessment of Virologic Failure
Description: •Assess the development of viral resistance in subjects experiencing virological failure
Time Frame: Within 48 weeks of randomization to study medications
Measure: Number; unit: participants with resistance for failure
Arm/Group | Once-daily Darunavir and Ritonavir | Twice-daily Darunavir and Ritonavir
Number analyzed (Participants) | 30 | 30
participants with resistance for failure | 0 | 0

6. Secondary Outcome: Number of Participants With Greater Than 95% Adherence at 48 Weeks
Description: Characterize adherence to once-daily versus twice-daily darunavir/ritonavir containing regimens using the Modified Medication Adherence Self-Report Inventory (M-MASRI) scale
Time Frame: Within 48 weeks of randomization to study medications
Population: Percentage of >95% adherence at week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Once-daily Darunavir and Ritonavir | Twice-daily Darunavir and Ritonavir
Number analyzed (Participants) | 27 | 27
Participants | 22 | 20

7. Secondary Outcome: Secondary Efficacy Endpoints
Description: •Proportion of subjects with plasma HIV-1 RNA <40 c/mL at Week 24
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Once-daily Darunavir and Ritonavir | Twice-daily Darunavir and Ritonavir
Number analyzed (Participants) | 30 | 30
Participants | 29 | 25

ADVERSE EVENTS:
Time Frame: 48 weeks during the trial, and 30 days after participant completion of the trial
Arm/Group | Once-daily Darunavir/Ritonavir | Twice-daily Darunavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The sample size was not adequately powered to evaluate non-inferiority, which might be clinically relevant. As a single-center study, identifying an appropriate number of eligible patients to determine non-inferiority was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No